CLINICAL TRIAL: NCT04338386
Title: Detection and Pathogenesis of Novel Protein F
Status: Not yet recruiting | Type: Observational
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YX-2020-B002
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Disease; Multiple Myeloma
Keywords: diagnosis; protein; cardiac disease; multiple myeloma; globulin
MeSH Terms: conditions — Heart Diseases; Multiple Myeloma; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From December 6, 2019 to March 23, 2020, the research group of Qingkun Fan found a novel protein(temporarily named protein F) in heparin anticoagulant plasma of three patients with heart disease. One patient was diagnosed with multiple myeloma.However, protein F cannot be detected by serum protein electrophoresis. Preliminary studies have shown that this novel protein F have an obvious absorption peak at about 600nm. Placed at 2-8 degrees for 7 days, protein F will be isolated from heparin plasma. To the naked eye, protein F appear to be transparent jelly between the red blood cells and the plasma. The specific protein F, how it is produced, how it causes disease are still unknown. This study will explore how to detect protein F and how it is produced.

DETAILED DESCRIPTION:
Protein F screening was performed on anticoagulant blood plasma with heparin Lithium or blood serum by in-house turbidimetric method in Automatic biochemical analyzer.

All patients were followed-up for 3 years by telephones, routine appointment out-patient clinic or returning visit.

ELIGIBILITY:
Inclusion Criteria:

* Testing total protein and albumin
* Testing routine blood test

Exclusion Criteria:

* high triglycerides (TG>5.00 mmol/L)
* hyperbilirubinemia (TBIL>170 mmol/L)
* fat emulsion used in past 3 days
* patients with hemolytic disease
* pregnant and lactating women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with heart diesease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2025-03-14 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Concentration of plasma protein F content | six month
  the protein F content was measured by turbidimetric assay in automatic biochemical analyzer

SECONDARY OUTCOMES:
Number of Participants with Multiple myeloma | 3 years
  Develop or be diagnosed with multiple myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlu Zhang, MD，Ph,D, Study Chair — Wuhan Asia Heart Hospital

IPD SHARING:
Plan to Share IPD: Undecided